CLINICAL TRIAL: NCT06778447
Title: Randomized, Sham-Controlled, Multi-Center, Double-Blind Clinical Trial Evaluating the Safety and Efficacy of Nucleus Pulposus Allograft to Supplement Nucleus Pulposus Tissue in Participants With Lumbar Discogenic Pain Associated With Degenerative Disc Disease
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of Nucleus Pulposus Allograft in Participants With Degenerative Disc Disease
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VIA-2024-002
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; Disc Degeneration; Lumbar Discogenic Pain
Keywords: Degenerative Disc Disease; Lumbar Discogenic Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Up to 496 subjects at up to 20 investigational sites in the United States.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIA Disc NP (Experimental): A single dose, intradiscal delivery of 100mg of VIA Disc NP mixed with sterile saline according to product Instructions for Use (IFU) and administered at up to two affected levels, L1-S1.
  Interventions: Other: VIA Disc NP
- Sham (Sham Comparator): The procedure will be identical to the investigational procedure with the following exception: A 20G spinal needle will be carefully inserted through the skin and muscle of the back but WILL NOT penetrate the annulus fibrosus of the intervertebral disc. No saline or VIA Disc NP will be injected.
  Interventions: Other: Sham

INTERVENTIONS:
Other: VIA Disc NP — VIA Disc NP is processed from donated cadaveric disc tissue, lyophilized, and micronized to particles.
  Other Names: VIA Disc Nucleus Pulposus Allograft
  Arms: VIA Disc NP
Other: Sham — A 20G spinal needle will be carefully inserted through the skin and muscle of the back but WILL NOT penetrate the annulus fibrosus of the intervertebral disc. No saline or VIA Disc NP will be injected.
  Arms: Sham

SUMMARY:
VIA Disc NP is a non-surgical intervention intended to supplement nucleus pulposus tissue in degenerated intervertebral discs.

This is a randomized, sham-controlled, multi-center, double-blind clinical trial with an open label roll-in period of one participant per site in which participants with lumbar discogenic pain associated with DDD will receive one VIA Disc NP treatment to each affected level (up to 2 levels). Participants enrolled after the roll-in stage will be randomized on a 2:1 basis to receive either a single VIA Disc NP intradiscal injection at 1 or 2 levels or the sham procedure at 1 or 2 levels. At 12 months, participants in the sham arm with continued symptoms may cross-over, receive VIA Disc NP, and will restart the study visit schedule, completing an additional 12 months of follow-up post-cross-over.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 to 85 years old
* Diagnosis of moderate to severe DDD on MRI, Modified Pfirrmann Grade 3-7
* Chronic axial midline low-back pain in the absence of lower extremity motor/sensory/reflex changes with or without referred non-radicular leg pain for at least 6 months prior to screening; unresponsive to at least 3 months of conservative care
* Low-back pain severity score of ≥ 40 to ≤ 90 mm on the VAS
* ODI score of ≥ 40 to ≤ 80
* Positive sustained hip flexion test
* Demonstrated intolerance to sitting
* Able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study
* Willing and able to comply with all study procedures and availability for the duration of the study with a life expectancy of > 2 years

Exclusion Criteria:

* Contraindications to the proposed sedation/anesthetic protocol
* Involvement of more than two lumbar discs as evidenced by 3 or more discs with Modified Pfirrmann grade of 3 or greater
* Disc height of less than 4mm for any disc between L1-S1
* Symptomatic vertebral compression fracture
* Previous surgical treatment of the lumbar spine
* History of sacroiliac (SI) joint fusion within the past six months
* Received lumbar epidural or intradiscal steroid injection, lumbar facet joint steroid injection, lumbar radiofrequency ablation, provocative or anesthetic discography, SI joint pain injection, injection of methylene blue, dextrose, glucosamine, and chondroitin sulfate, or biacuplasty within 3 months of the Day 0 procedure
* Received intraosseous radiofrequency nerve ablation procedure at the same or adjacent level (e.g., Basivertebral nerve ablation or sinuvertebral nerve ablations)
* Received prior intradiscal stem cell/progenitor cell therapy or other biological intervention (e.g., MSC, PRP) at the target level within 12 months of the Day 0 procedure
* Evidence of dynamic instability on lumbar flexion-extension radiographs (>3 mm)
* Grade 2 or higher spondylolisthesis at the target level, lumbar spondylitis or other undifferentiated spondyloarthropathy, or Type III Modic changes adjacent to the target disc
* Radiographic evidence of a full thickness annular tear at the target disc or other abnormal disc morphology
* Clinical suspicion of facet pain as primary pain generator
* A systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study (e.g. current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, recent history of myocardial infarction, uncontrolled diabetes (>7.0% HbA1C), etc.)
* Received VIA Disc NP previously.
* Deemed unsuitable for clinical study participation by the Investigator
* Evidence of substance abuse (including marijuana); note: subjects using prescribed extended-release narcotics (e.g., fentanyl patch, MS Contin, oxycontin) within the 3 months prior to screening and subjects on long-acting opioids may be given option to wean off opiates before enrollment; subjects on short-acting opiates (e.g., hydrocodone, oxycodone, tramadol, etc.) may be included and utilization monitored after the treatment
* Opioid use of more than 90 MME/day
* Currently receiving treatment with radiation, chemotherapy, immunosuppression, or chronic steroid therapy (prednisone, or its equivalent, use of up to 5 mg/qd, or inhalation steroids for asthma is allowed)
* Metal or ceramic implants in the lumbar spine region
* Contraindications to MRI, including non-MRI compatible devices and active implantable devices such as spinal cord stimulators, intrathecal pumps, etc.
* Involved in ongoing or closed (within 6 months of screening visit) litigation related to their back pain condition
* Any mental instability, unstable bipolar disorders, unmanaged post-traumatic stress disorder (PTSD) or uncontrolled anxiety/depression and/or require new or changed anti-depressants or anti-psychotic medications within 3 months of enrollment
* Diagnosis of any traumatic neurological disorders that may impact the study as per the judgement of the Investigator
* Women who are pregnant or breastfeeding at the time of enrollment and/or plan to become pregnant during the study; pregnancy is confirmed by:
* a positive pregnancy test during the screening visit
* self-reported pregnancy
* Women of childbearing potential (WOCBP) who are not using a reliable form of contraception (as determined by the Investigator)
* Received any experimental drug or device to treat the same condition used within 6 months prior to the screening visit or during the course of the clinical trial
* Other persistent pain/nerve issues including, for example, radiculopathy, leg pain, cauda equine syndrome, etc.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Proportion of participants achieving MCID in VAS score from baseline to 12 months. | Baseline to 12 Months
  The primary efficacy endpoint is the proportion of participants who achieve a minimal clinically important difference (MCID), defined as at least a 30% reduction in back pain VAS score from baseline to 12 months, in the VIA Disc NP group compared to that in the sham-control group.
Primary Safety Endpoint - Proportion of participants reporting treatment-related AEs at 12 months. | Baseline to 12 Months
  The primary safety endpoint will be the proportion of participants that experience one or more treatment-related (Investigational Product (IP) or procedure), adverse events (AE) in the VIA Disc NP group compared to the sham-control group at 12 months.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Interventional Pain Management Napa Valley Orthopedic Medical Group, Napa, California
  - Source Healthcare, Santa Monica, California
  - Premier Spine and Pain Institute, Thornton, Colorado
  - The Orthopaedic Institute, Gainesville, Florida
  - Georgia Pain Management, Woodstock, Georgia
  - Henry Community Health, New Castle, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Paradigm Health System, Slidell, Louisiana
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Crystal Coast Pain Management, New Bern, North Carolina
  - Pacific Sports & Spine, Eugene, Oregon
  - Pain Specialists of America, Killeen, Texas
  - Procura Pain & Spine, Shenandoah, Texas
  - Precision Spine Care, Tyler, Texas
  - The Spine and Nerve Center C/O Clinical Research, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No